CLINICAL TRIAL: NCT05772351
Title: Preoperative Micronized Flavonoid Fraction (MFF) Use in Multimodal Anesthesia in Anorectal Surgery: Study Protocol for Prospective, Randomized, Placebo-controlled, Double-blind Study
Brief Title: Preoperative Micronized Flavonoid Fraction (MFF) Use in Multimodal Anesthesia in Anorectal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center of Endourology "Endocenter" (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5995465475
Record Dates: First submitted 2023-03-06; First posted 2023-03-16 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Hemorrhoids; Hemorrhoid Pain; Hemorrhoidal Bleeding
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): Patients of the experimental group received Detralex® 1000 mg QD for 15 days before the operation, 3000 mg starting from day 1 after the surgery for 4 days, then 2000 mg for the next 3 days and 1000 mg till day 30 after surgery
  Interventions: Drug: micronized flavonoid fraction
- Control group (No Intervention): Patients of the control group received a tablet containing starch.

INTERVENTIONS:
Drug: micronized flavonoid fraction — Patients of the experimental group received Detralex® 1000 mg QD for 15 days before the operation, 3000 mg starting from day 1 after the surgery for 4 days, then 2000 mg for the next 3 days and 1000 mg till day 30 after surgery.
  Under spinal anesthesia appropriate surgical intervention was performed. After the surgery, the patient was given a questionnaire and a scale for assessing pain at rest and during defecation within the first 2 weeks after surgery. During the hospital stay, the nurse filled out a section on the drugs used; after discharge, the patient filled out this section for 7 days after the surgery. After 30 days, the side effects section was filled out, and the quality of life was assessed on days 7 and 30. Also, the patients indicated in a separate column on which day after the surgery they were able to return to normal living or go to work.
  Arms: Experimental group

SUMMARY:
Aim: To assess the efficiency of the micro-flavonoid fraction (MMF) administration prior to anorectal surgery with spinal anesthesia on postoperative pain severity reduction.

Methods: Patients who meet the following criteria are included: participants must be diagnosed with surgical treatment of anorectal diseases. All participants are randomly divided into 2 groups: the first one gets a tablet with 1000 mg MFF (Detralex®), the second one gets a tablet containing starch per os 14 days before surgery (72 participants per arm). Then patients of each group will continue MFF administration for 30 days after surgery. Patients of both arms receive spinal anesthesia and undergo surgery. Following the procedure the primary and secondary outcomes are evaluated: frequency of the opioid drugs intake, the severity of the postoperative pain syndrome, duration and frequency of other drugs intake, readmission rate, overall quality of life, time from the procedure to returning to work and the complications rate, C-reactive protein level.

Discussion: the MFF intake allows reducing the severity of the hemorrhoidal disease symptoms during conservative treatment. In addition, the Detralex® efficacy has been proven in postoperative pain reduction for patients diagnosed with varicose veins of the lower extremities. The investigators intend to evaluate the feasibility of the preoperative MFF administration for the postoperative pain reduction and the decrease of the postoperative complications in patients with hemorrhoidal disease.

ELIGIBILITY:
Inclusion Criteria:

* Stage 2-4 hemorrhoidal disease;
* Presence of indications for elective surgery (open hemorrhoidectomy) using mono or bipolar coagulation possibly combined with other minimally invasive methods: hemorrhoidopexy and mucopexy, Ligasure hemorrhoidectomy;
* Absence of other diseases that cause pain;
* Class I, II ASA anesthesia risk;

Exclusion Criteria:

* The presence of the following diseases: paraproctitis, inflammatory bowel disease, metabolic or endocrine disorders, alcoholism, drug use, blood clotting disorders, and history of diseases in the anorectal region;
* Contraindicated or technically impossible subarachnoid anesthesia;
* Patients who refused to participate;
* Pregnant women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2021-11-25 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
rate of prescribing opioid analgesics | 7 days after surgery
  the rate of prescribing opioid analgesics to prevent the pain from rising above VAS 5 after surgery

SECONDARY OUTCOMES:
pain at rest and during defecation | 15 days after surgery
  The pain was assessed using a visual analogue scale (VAS, 0 to 10 points, where 10 is the maximum score).
other medications use | 7 days after surgery
  the need for other medications after surgery
readmission rate | 30 days after surgery
The life quality rate | 7 and 30 days
  The overall quality of life was assessed using the EQ-5D patient questionnaire.
time from surgery to return to work | during 30 days after surgery
complication rates | within 30 days after the procedure
  bleeding, urinary retention, infectious complications

CONTACTS AND LOCATIONS:
Locations (1):
- Lomonosov Moscow State University, Fundamental Medicine Faculty, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No